CLINICAL TRIAL: NCT01882699
Title: A Multi-center, Prospective, Non-randomized Study to Determine Durability of Effectiveness of the Cerêve Sleep System Following 30 Days in Home Use and Home Use Patterns Over 6 Months
Brief Title: 30 Days in Home Use and Home Use Patterns Over 6 Months
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cereve, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP-004
Record Dates: First submitted 2013-05-30; First posted 2013-06-20 (Estimated); Last update posted 2015-05-22 (Estimated); Status verified 2015-05

CONDITIONS: Primary Insomnia
Keywords: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cereve sleep system (Experimental): Cereve sleep system
  Interventions: Device: Cereve Sleep System

INTERVENTIONS:
Device: Cereve Sleep System — cerebral hypothermia

SUMMARY:
This study will build upon a previously approved protocol entitled "A multi-center prospective, blinded, randomized crossover study to compare the Cerêve Sleep System at two different temperatures in primary insomnia patients" (CIP-003; CER1-01-090). In that study, 150 insomnia patients were targeted to be randomized to complete in lab assessments of sleep using the Cerêve Sleep System. In this follow-on study, 36 patients who completed the in lab study will be enrolled to complete 2 phases of in home use of the device. In the first phase, the durability study, 30 patients are targeted to complete additional in lab assessments following 30 days of in home use of the device. In the second phase, the home use pattern study, 24 patients are targeted to complete an additional 5 months of in home use in which their use patterns will be monitored.

Hypothesis:

EEG sleep latency and sleep efficiency following 30 days in home use of the device at 14-16°C will be similar to those measures after the initial acute, 2-night use in the parent study in the 14-16°C condition. The device will demonstrate a benign safety profile over 6 months in home use.

DETAILED DESCRIPTION:
Study Design Objectives of the Clinical Investigation

* Assess polysomnographically measured sleep latency and sleep efficiency following 30 days in home use of the device and compare these measures with those following initial in lab use in the CIP-003 protocol.
* Determine the long-term use patterns of the Cerêve Sleep System in the environment of intended use.

Study Design Overview A multi-center, prospective, non-randomized, two phase study to determine durability of effects following 30 days of in home use (phase I) and home use patterns over an additional 5 months in home use of the Cerêve Sleep System (phase II).

A total of 30 evaluable subjects will be targeted to complete phase I and a total of 24 evaluable subjects will be targeted to complete phase II. It is anticipated that 36 subjects will be enrolled into the CIP-004 protocol to obtain the numbers of evaluable subjects described.

During in home use in both the durability phase and the home use patterns phase, the subject will be asked to use the device for a minimum of three nights each week for at least 4 hours on each of these nights up to seven nights each week. Subjects will complete a weekly home use log throughout both phases of the study.

ELIGIBILITY:
Inclusion Criteria:

* Must have completed the in-lab protocol CIP-003 and have signed an informed consent to participate in this follow-on study.
* Sleep latency and sleep efficiency data are available from the 2 in-lab PSG nights from CIP-003 in the 14-16° condition, as confirmed by the core laboratory.

Exclusion Criteria:

* Use of medications known to affect sleep or wake function (e.g., hypnotics, benzodiazepines, antidepressants, anxiolytics, antipsychotics, antihistamines, decongestants, beta blockers, corticosteroids) are excluded for the durability phase, through the in-lab studies, in this protocol; Beta blockers which do NOT cross the blood brain barrier are acceptable.
* Consumption of more than one alcoholic drinks per day, or more than 7 drinks per week prior to study entry and during the durability phase, through the in-lab studies, in this protocol.
* Caffeinated beverages > 4/day or the equivalent of more than 4 cups of coffee during the durability phase, through the in-lab studies, in this protocol.
* Unable to read or understand English

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-05; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
sleep latency | 30 days
  latency from time in bed to persistent sleep
sleep efficiency | 1 month
  time asleep/time in bed

CONTACTS AND LOCATIONS:
Overall Officials: Alan Lankford, PhD, Principal Investigator — Sleep Center of Georgia; David Mayleben, PhD, Principal Investigator — Community Research; Neil Feldman, MD, Principal Investigator — Clinical Research Group of St. Petersburg; Russell Rosenberg, PhD, Principal Investigator — Neurotrials
Locations (4):
- United States (4):
  - Neil Feldman, Saint Petersburgh, Florida
  - Alan Lankford, Atlanta, Georgia
  - Russell Rosenberg, Atlanta, Georgia
  - David Mayleben, Crestview Hills, Kentucky